CLINICAL TRIAL: NCT04077944
Title: Maternal Serum Levels of Selected Trace Elements and Heavy Metals in Pregnancies Complicated With Preterm Prelabor Rupture of Membranes
Brief Title: Trace Elements and Heavy Metals at PPROM
Acronym: metals&PROM
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH4
Record Dates: First submitted 2019-08-31; First posted 2019-09-04 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Preterm Rupture of Membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm prelabor rupture of membranes: The diagnosis of Preterm prelabor rupture of membranes was made in the case of apparent spontaneous leakage of AF from the cervical canal during sterile speculum inspection before the onset of active labor at 37 weeks of pregnancy. The study population consisted of 55 women with a singleton pregnancy who were diagnosed with pP-ROM between 24+0 and 36+6 weeks of gestation.
  The Amnisure test (AmniSure International LLC, Boston, MA) was used when there was inconclusive results to confirm the final diagnosis. The gestational age was determined by calculation from the last menstrual period and supported by the ultrasonography measurements at the first trimester of gestation.
  Interventions: Diagnostic Test: maternal serum concentration of trace elements and heavy metals levels
- Control: The control cases were recruited from the healthy pregnant women with a gestational age-matched cohort who admitted for routine obstetric care to our outpatient clinic. Sixty healthy pregnant women who delivered at term were included in the study as the control group.
  Interventions: Diagnostic Test: maternal serum concentration of trace elements and heavy metals levels

INTERVENTIONS:
Diagnostic Test: maternal serum concentration of trace elements and heavy metals levels — The maternal serum levels of trace elements and heavy metals in both groups were measured using an inductively coupled plasma-mass spectrometry (ICP-MS)

SUMMARY:
Objectives: To evaluate maternal serum trace elements and heavy metals namely, aluminum (Al), chromium (Cr), manganese (Mn), cobalt (Co), nickel (Ni), copper (Cu), zinc (Zn), arsenic (As), molybdenum (Mo), cadmium (Cd), tin (Sn), antimony (Sb), mercury (Hg), and lead (Pb) in pregnant women complicated by preterm prelabour rupture of the membranes (pP-ROM) and to compare the results with healthy pregnancies.

Methods: Maternal serum levels of Al, Cr, Mn, Co, Ni, Cu, Zn, As, Mo, Cd, Sn, Sb, Hg, and Pb were measured in the study group, which included 55 pregnant women complicated with pP-ROM and 60 healthy pregnancies (control group) with respect to maternal age and gestational weeks. The maternal serum levels of trace elements and heavy metals in both groups were measured using an inductively coupled plasma-mass spectrometry (ICP-MS) and compared.

DETAILED DESCRIPTION:
This current observational study was conducted at Cengiz Gokcek Women's and Children's Hospital Gaziantep, Turkey at the Department of Obstetrics and Gynecology between dates of August 2018 and March 2019. The experiment was conducted according to the Declaration of Helsinki. All subjects included in the study gave oral and written informed consents. The study population consisted of 55 women with a singleton pregnancy who were diagnosed with pP-ROM between 24+0 and 36+6 weeks of gestation. The control cases were recruited from the healthy pregnant women with a gestational age-matched cohort who admitted for routine obstetric care to our outpatient clinic. Sixty healthy pregnant women who delivered at term were included in the study as the control group. All patients will gave their oral and written informed consent before their inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* preterm prelabor rupture of the membranes
* healthy pregnancy

Exclusion Criteria:

* • pregnant women who had the diagnosis of chorioamnionitis at the time of first admission

  * women with chronic medical diseases
  * gestational diabetes mellitus
  * women with a history of drug use throughout pregnancy
  * drug users
  * pregnant women who have received any treatment for pP-ROM at the time of admission
  * patients who had fetal congenital abnormalities or genetic syndromes
  * genetic syndromes
  * multiple gestation
  * active labor
  * fetal hypoxia
  * fetal growth restriction

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — preterm prelabour rupture of the membranes is described as rupture of the amniotic membranes prior to 37 weeks of completed gestation.
Study Population: The investigators consecutively will recruite 55 subjects with preterm prelabor rupture of the membranes, and 60 healthy preganancies will selected for the control group.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint | 3 months
  The primary endpoint in this analysis is to evaluate maternal serum trace elements and heavy metals namely, aluminum (Al), chromium (Cr), manganese (Mn), cobalt (Co), nickel (Ni), copper (Cu), zinc (Zn), arsenic (As), molybdenum (Mo), cadmium (Cd), tin (Sn), antimony (Sb), mercury (Hg), and lead (Pb) in pregnant women complicated by preterm prelabor rupture of the membranes (pP-ROM) and to compare the results with healthy pregnancies.
  The elements, Al, Cr, Mn, Co, Ni, Cu, Zn, As, Mo, Cd, Sn, Sb, Hg and Pb were measured using an inductively coupled plasma-mass spectrometry (ICP-MS) (Thermo Scientific ICAPQc, USA).
  In the present study, only the maternal serum levels of fourteen different TEs and HMs were evaluated in order to examine the association between the occurrence of pP-ROM and these elements.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Igbinosa I, Moore FA 3rd, Johnson C, Block JE. Comparison of rapid immunoassays for rupture of fetal membranes. BMC Pregnancy Childbirth. 2017 Apr 26;17(1):128. doi: 10.1186/s12884-017-1311-y. PMID 28446135
- [Background] Wang KC, Lee WL, Wang PH. Early and late preterm premature rupture of membranes. J Chin Med Assoc. 2017 Oct;80(10):613-614. doi: 10.1016/j.jcma.2017.03.006. Epub 2017 May 2. No abstract available. PMID 28476444
- [Result] Vigeh M, Yokoyama K, Shinohara A, Afshinrokh M, Yunesian M. Early pregnancy blood lead levels and the risk of premature rupture of the membranes. Reprod Toxicol. 2010 Nov;30(3):477-80. doi: 10.1016/j.reprotox.2010.05.007. Epub 2010 May 16. PMID 20576532

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT04077944/SAP_000.pdf